CLINICAL TRIAL: NCT01535703
Title: Comparison of Cardiac Output Measurement Between Invasive Method (Transpulmonary Thermodilution) and Non Invasive Method (Photoplethysmography) : an Observational Study
Brief Title: Comparison of Cardiac Output Measurement Between Transpulmonary Thermodilution and Photoplethysmography
Acronym: PANEX
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 11-007
Record Dates: First submitted 2012-02-07; First posted 2012-02-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Monitoring could secure management for patient but stay invasive. The purpose of this study was to compare,after cardiac surgery, the cardiac output measurement between transpulmonary thermodilution(reference method) and digital photoplethysmography (non invasive) for absolute value and dynamics changes before and after fluid expansion for patients with indication of fluid challenge.

DETAILED DESCRIPTION:
* The time frame of the study period was included between the arrival at the ICU after cardiac surgery and before spontaneous breathing on mechanical ventilation
* Time-to-event outcome measures was period of time between the arrival at the ICU after cardiac surgery and before spontaneous breathing on mechanical ventilation. The event (hypotension) was defined as systolic arterial pressure under 90mmHg,less than 40mmHg, mean arterial pressure under 70mmHg, tachycardia upper 100 beats/min, presence of skin mottling, low cardiac output or previous blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Postcardiac surgery patients with arterial pressure monitoring and transpulmonary thermodilution monitoring with indication of fluid challenge
* Patients more than 18 years old

Exclusion Criteria:

* Patients under 18 years old
* Pregnant women
* Patient without invasive monitoring
* Urgency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post cardiac surgery intensive care patients with arterial pressure monitoring and transpulmonary thermodilution monitoring with indication of fluid challenge.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Correlation, percentage error, bias, precision and limits of agreement for change in cardiac output measured by digital photoplethysmography compared with transpulmonary thermodilution during fluid expansion | During admission in ICU after cardiac surgery and before spontaneous breathing-measurements will be complete within 60 minutes of starting fluid expansion
  Analysis of correlation, percentage error, bias, precision and limits of agreement for change in cardiac output measured by digital photoplethysmography compared with transpulmonary thermodilution during fluid expansion

SECONDARY OUTCOMES:
Bias and limits of agreement for change in arterial pressure measured by digital photoplethysmography compared with intra radial artery catheter during volume expansion | During admission in ICU after cardiac surgery and before spontaneous breathing-measurements will be complete within 60 minutes of starting fluid expansion
  Analysis of agreement, bias and precision between arterial pressure from digital photoplethysmography and intra radial artery catheter
Predictive value of fluid responsiveness by the variation of pulse pressure variation measuring by radial artery catheter and digital photoplethysmography | During admission in ICU after cardiac surgery and before spontaneous breathing-measurements will be complete within 60 minutes of starting fluid expansion
  Analysis of the predictive value of fluid responsiveness with AUC receiving operating curve by the variation of pulse pressure variation measuring by radial artery catheter and digital photoplethysmography
Predictive value of fluid responsiveness by three different localisation of plethysmographic variability index sensor: forehead, digital and ear position | During admission in ICU after cardiac surgery and before spontaneous breathing-measurements will be complete within 60 minutes of starting fluid expansion
  Analysis of the predictive value of fluid responsiveness with AUC receiving operating curve for each localisation of sensor of plethysmography variability index

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Olivier Fischer, M.D., Principal Investigator — University Hospital, Caen
Locations (1):
- University Hospital, Caen, Caen, France